CLINICAL TRIAL: NCT06744933
Title: Self-administered Auricular Acupressure Integrated With a Smartphone Application for Weight Reduction in Patients With Obesity Accompanied With Obesity-related Comorbid Illness: A Randomised Controlled Clinical Trial
Brief Title: Auricular Acupressure Integrated With a Smartphone Application for Weight Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Collaborators: Hospital Authority Hong Kong West Cluster (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-04-75-CMDF240401
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Obesity and Metabolic Syndrome
Keywords: auricular acupressure; auricular therapy; weight reduction; obesity; metabolic syndrome; mobile health; mHealth; smartphone application; traditional Chinese medicine; TCM; ear acupressure; weight loss
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-administered auricular acupressure integrated with a smartphone application (Experimental): Patients in this group will undergo TCM syndrome differentiation, and then be given 6 to 8 hypoallergic Vaccariae Semen ear patches on one ear. 6 of the auricular acupoints will be compulsory, while the additional 1 to 2 acupoints will be selected according to the TCM syndrome of the patient. These 6 mandatory acupoints were selected according to previous literature and expert opinion. The research staff will use an ear model to demonstrate to the patients how to press on the auricular acupoints and require them to perform a return demonstration to ensure they can perform auricular acupressure correctly by themselves. The patient will then be required to visit the clinic twice a week and will change a new set of ear patches on the same acupoints of the opposite ear. This intervention will last for 8 weeks. Their BMI (and weight) and their satiety level will be monitored once a week while they visit the clinic.
  Interventions: Combination Product: Self-administered auricular acupressure integrated with a smartphone application
- Usual care (No Intervention): The usual care group will receive no intervention. They will only be assessed on the outcomes.

INTERVENTIONS:
Combination Product: Self-administered auricular acupressure integrated with a smartphone application — 6 to 8 Vaccariae Semen ear patches will be affixed on one ear of the patient. The patient will be required to press on the ear patches 3 times a day, and 30 minutes before a meal. Every 3 to 4 days, the patient will visit the clinic to change a new set of ear patches on the same auricular acupoints of the opposite ear alternately. The whole course of intervention will be 8 weeks. The smartphone app will send scheduled pop-up notifications to remind patients to press on the ear patches. The patient will be required to enter the number of times pressing and of defaecation every day on the smartphone application. The smartphone application will send more notifications to the patient if he/ she has a low compliance. When the participants record the number of times pressing on the auricular acupoints, positive reinforcement messages will pop-up, such as "Excellent job!" for those with good compliance while "You are almost there! Keep going!" for those with poor compliance.
  Arms: Self-administered auricular acupressure integrated with a smartphone application

SUMMARY:
The goal of this clinical trial is to learn whether self-administered auricular acupressure integrated with a smartphone application works to reduce weight in patients with obesity accompanied with obesity-related comorbid illness. The main questions it aims to answer are:

* Is there significant difference in the Body Mass Index (BMI) between the self-administered auricular acupressure integrated with a smartphone app (Version 2) group (experimental group) and the usual care group, in people with obesity accompanied with metabolic syndrome?
* Are there significant differences in other anthropometric parameters between the two groups? These parameters include waist circumference, body fat percentage, skeletal muscle percentage, and waist-to-hip ratio.
* Are there any significant differences in obesity-related parameters between the two groups? These parameters include blood lipid profile (triglyceride, total cholesterol, low-density lipoprotein (LDL), and high-density lipoprotein (HDL)), blood glucose concentrations (fasting glucose and glycated haemoglobin/ HbA1c), and blood pressure.

Participants in the experimental group will:

* Be affixed with 6 to 8 hypoallergic Vaccariae Semen ear patches on one ear each time
* Visit the clinic twice a week to change a new set of ear patches on the opposite ear
* Will undergo this intervention for 8 weeks
* Install a smartphone application which will send pop-up notifications to remind them to press on the ear patches regularly every day
* Keep a record on the number of times pressing on the smartphone application

DETAILED DESCRIPTION:
Obesity has become a global public health problem, and its prevalence is surging in Asia. According to the Population Health Survey in 2020-22 by the Department of Health in Hong Kong, over 50% of Hong Kong general population was classified as obese (Body Mass Index (BMI) ≥ 25.0 kg/m2) or overweight (BMI ≥ 23.0 kg/m2), and central obesity was accounting for 37.8%. As the population ages, overweight and obesity become more and more serious. The incidence of metabolic syndrome is increasing yearly around the world. According to the health survey mentioned above, the prevalence of various disorders that constitute metabolic syndrome ranged from 8.5% (hyperglycaemia or diabetes) to 51.9% (raised blood cholesterol or hypercholesterolaemia). Metabolic syndrome is a collective disorder comprising abdominal obesity, abnormal blood sugar, dyslipidaemia and hypertension, which seriously affects the health of the body and cannot be ignored.

Western medications currently used for weight reduction include centrally-acting appetite suppressants, blockers inhibiting intestinal fat absorption, and metabolic stimulants. Although these Western medications are effective in treating obesity, the associated adverse effects limit their clinical applications. Long-term use of weight reduction medications can cause many adverse effects in the cardiovascular system, digestive system, and liver. Bariatric surgery, such as gastric bypass or sleeve gastrectomy, may cause serious complications, for instance, bleeding, intestinal obstruction, anorexia, or gastric perforation.

In recent years, mobile health (mHealth) has played an essential role in preventing and managing chronic diseases. In the fields of both medicine and nursing care, smartphone apps are widely used to assist in the intervention of chronic diseases. A smartphone app can remind participants to press the ear patches promptly and correctly to achieve optimum treatment effect. In addition, the smartphone app can also provide relevant health information to encourage people with obesity to change their unhealthy lifestyles.

Through literature review and expert consultation, the research team selected six auricular acupoints that were found to have specific effects on weight reduction, namely Shenmen, Stomach, Endocrine, External nose (also known as "hunger point"), Large intestine, and Forehead. Not only does the smartphone app remind the participants to press on the auricular acupoints, the participants can also learn about the benefits of auricular acupressure, the locations of auricular acupoints, and the correct way of executing auricular acupressure on the smartphone app.

This proposed research project aims to evaluate the efficacy of self-administered auricular acupressure integrated with a smartphone app (Version 2), a composite intervention for people with obesity accompanied with metabolic syndrome. It will be a two-arm randomised clinical trial conducted in a community setting.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. Body Mass Index (BMI) ≥ 30 kg/m2 and /or abdominal obesity (i.e., central obesity), that is, male waist circumference ≥ 90cm while female waist circumference ≥ 80cm;
3. fulfils diagnostic criteria for metabolic syndrome with any two or more of the following: (a) blood pressure ≥ 130/85 mmHg and/ or confirmed diagnosis of hypertension with treatment; (b) fasting blood glucose ≥ 100 mg/dl (5.6 mmol/L) and/ or confirmed diagnosis of diabetes with treatment; (c) fasting triglyceride ≥ 150 mg/dl (1.7 mmol/L) and/ or received specific treatment on dyslipidaemia; (d) fasting high-density lipoprotein (HDL) < 40mg/dl (< 1.03mmol/L) in male; < 50mg/dl (< 1.29 mmol/L) and/ or received specific treatment on dyslipidaemia; These standards are based on the diagnostic criteria for metabolic syndrome from the World Health Organisation (1999), the International Diabetes Federation Criteria (2005), and the Chinese Diabetes Society (2000);
4. are taking medications and receiving follow-up medical consultation [Note: With the consent of the participants, the researchers (i.e., the RCA and the RA) will verify relevant medical records in the follow-up appointments];
5. taken no weight control measures in the past 6 months;
6. has no trauma, inflammation or pathological lesion on ears;
7. is a smartphone user.

Exclusion Criteria:

1. has any eating disorder (screened by the 5-item SCOFF questionnaire);
2. has drug-induced obesity;
3. is pregnant;
4. has cognitive impairment (Abbreviated Mental Test (Hong Kong version), AMT score below 6 (less than or equal to 5) will be excluded.);
5. has cancer; or
6. has a severe body disability, such as hemiplegia, that may prevent following instructions to use the smartphone.
7. is planning to have weight-reduction treatment(s) (such as medications targeted for weight reduction, and bariatric surgery) in the coming 6 months.
8. is taking the following medications that potentially affect the body weight:

   * Corticosteroids (e.g., prednisone and dexamethasone)
   * Second generation antipsychotics (e.g., olanzapine, clozapine, quetiapine and risperidone)
   * Levothyroxine
   * FDA-approved medications for obesity or weight loss (e.g., phentermine, diethylpropion, phendimetrazine, phentermine + topiramate extended release (ER), naltrexone + bupropion ER, orlistat, liraglutide, semaglutide and GLP-1 (liraglutide/ semaglutide) + tirzepatide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-04-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in the mean Body Mass Index (BMI) at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  BMI is a continuous numerical scale. Zero is equivalent to no change in weight; Positive change is equivalent to weight gain; Negative change is equivalent to weight reduction.

SECONDARY OUTCOMES:
Change from baseline in mean waist circumference at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  Waist circumference is continuous numerical scale. Waist circumference will be measured midway between the edge of the lower ribs and the iliac crest. To ensure accuracy, each measurement will be taken twice and the average will be calculated. Zero is equivalent to no change. Broadly speaking, positive changes refer to unhealthy change and negative changes refer to healthy change.
Changes from baseline in mean body fat percentage and skeletal muscle percentage at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  They are all continuous numerical scales with reference ranges indicating a healthy state. Any value outside these reference ranges can be regarded as unhealthy. Body fat percentage and skeletal muscle percentage will be measured by Tanita BC-545N. For both of them, zero is equivalent to no change. Broadly speaking, for body fat percentage, positive changes refer to unhealthy change and negative changes refer to healthy change. Alternatively, for skeletal muscle percentage, positive change refers to healthy change and negative change refers to unhealthy change.
Change from baseline in mean waist-to-hip ratio at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  Waist-to-hip ratio is all continuous numerical scale. Waist and hip circumferences will be measured by hand. Zero is equivalent to no change. Positive change refers to a more apple-shaped body shape and negative change refers to a more pear-shaped body shape.
Changes from the baseline in the mean blood lipid profile at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  Blood lipid profile include triglyceride , total cholesterol, low-density lipoprotein (LDL) and high-density lipoprotein (HDL).They are all continuous numerical scales with reference ranges indicating a healthy state. Any value outside these reference ranges can be regarded as unhealthy. Zero is equivalent to no change. These parameters mainly measure the changes in patients with dyslipidaemia. As a result, positive changes in triglyceride, total cholesterol and LDL refer to unhealthy change and negative changes refer to healthy change. Positive change in HDL refers to healthy change and negative change refers to unhealthy change.
Changes from the baseline in the mean blood glucose concentrations at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  Blood glucose concentrations include fasting glucose and glycated haemoglobin/ HbA1c. They are all continuous numerical scales with reference ranges indicating a healthy state. Any value outside these reference ranges can be regarded as unhealthy. Zero is equivalent to no change. These parameters mainly measure changes in patients with diabetes. As a result, positive changes in fasting glucose and HbA1c refer to unhealthy change and negative changes refer to healthy change.
Change from the baseline in the mean blood pressure at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  Blood pressure is a continuous numerical scale. It mainly measures changes in patients with hypertension. As a result, positive changes in blood pressure (systolic and diastolic) refer to unhealthy change and negative changes refer to healthy change.
Differences in the change from baseline in BMI (and other parameters in the secondary outcomes) in patients in the experimental group with different TCM syndromes at one month and four months after the completion of the intervention | Baseline, one month post-intervention, and four months post-intervention
  TCM syndrome differentiation will be performed in patients in the experimental group. They will be classified into "Excessive", "Deficient", or "Deficiency-Excess Complex". Possible sub-classification may be performed. The changes in all outcome parameters (including primary and secondary outcomes) mentioned above will be compared across patients with different syndromes. Any significant difference detected among these syndromes may indicate positive or negative effect on a specific TCM syndrome type(s).

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Risk Assessment & Management Clinic, Tsan Yuk Hospital, Hong Kong
  - Sai Ying Pun Jockey Club General Out-patient Clinic, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ling J, Chen S, Zahry NR, Kao TA. Economic burden of childhood overweight and obesity: A systematic review and meta-analysis. Obes Rev. 2023 Feb;24(2):e13535. doi: 10.1111/obr.13535. Epub 2022 Nov 27. PMID 36437105
- [Background] Hsu CH, Wang CJ, Hwang KC, Lee TY, Chou P, Chang HH. The effect of auricular acupuncture in obese women: a randomized controlled trial. J Womens Health (Larchmt). 2009 Jun;18(6):813-8. doi: 10.1089/jwh.2008.1005. PMID 19445642
- [Background] Hsieh CH, Su TJ, Fang YW, Chou PH. Efficacy of two different materials used in auricular acupressure on weight reduction and abdominal obesity. Am J Chin Med. 2012;40(4):713-20. doi: 10.1142/S0192415X1250053X. PMID 22809026
- [Background] Hsieh CH, Su TJ, Fang YW, Chou PH. Effects of auricular acupressure on weight reduction and abdominal obesity in Asian young adults: a randomized controlled trial. Am J Chin Med. 2011;39(3):433-40. doi: 10.1142/S0192415X11008932. PMID 21598412
- [Background] Suen L, Wang W, Cheng KKY, Chua MCH, Yeung JWF, Koh WK, Yeung SKW, Ho JYS. Self-Administered Auricular Acupressure Integrated With a Smartphone App for Weight Reduction: Randomized Feasibility Trial. JMIR Mhealth Uhealth. 2019 May 29;7(5):e14386. doi: 10.2196/14386. PMID 31144666
- [Background] Granado-Font E, Flores-Mateo G, Sorli-Aguilar M, Montana-Carreras X, Ferre-Grau C, Barrera-Uriarte ML, Oriol-Colominas E, Rey-Renones C, Caules I, Satue-Gracia EM; OBSBIT Study Group. Effectiveness of a Smartphone application and wearable device for weight loss in overweight or obese primary care patients: protocol for a randomised controlled trial. BMC Public Health. 2015 Jun 4;15:531. doi: 10.1186/s12889-015-1845-8. PMID 26041131
- [Background] Eisenhauer CM, Hageman PA, Rowland S, Becker BJ, Barnason SA, Pullen CH. Acceptability of mHealth Technology for Self-Monitoring Eating and Activity among Rural Men. Public Health Nurs. 2017 Mar;34(2):138-146. doi: 10.1111/phn.12297. Epub 2016 Oct 18. PMID 27757986
- [Background] Semper HM, Povey R, Clark-Carter D. A systematic review of the effectiveness of smartphone applications that encourage dietary self-regulatory strategies for weight loss in overweight and obese adults. Obes Rev. 2016 Sep;17(9):895-906. doi: 10.1111/obr.12428. Epub 2016 May 18. PMID 27192162
- [Background] Lim R, Beekley A, Johnson DC, Davis KA. Early and late complications of bariatric operation. Trauma Surg Acute Care Open. 2018 Oct 9;3(1):e000219. doi: 10.1136/tsaco-2018-000219. eCollection 2018. PMID 30402562
- [Background] Chang SH, Stoll CR, Song J, Varela JE, Eagon CJ, Colditz GA. The effectiveness and risks of bariatric surgery: an updated systematic review and meta-analysis, 2003-2012. JAMA Surg. 2014 Mar;149(3):275-87. doi: 10.1001/jamasurg.2013.3654. PMID 24352617
- [Background] Wadden TA, Webb VL, Moran CH, Bailer BA. Lifestyle modification for obesity: new developments in diet, physical activity, and behavior therapy. Circulation. 2012 Mar 6;125(9):1157-70. doi: 10.1161/CIRCULATIONAHA.111.039453. No abstract available. PMID 22392863
- [Background] Ko GT. The cost of obesity in Hong Kong. Obes Rev. 2008 Mar;9 Suppl 1:74-7. doi: 10.1111/j.1467-789X.2007.00442.x. PMID 18307703
- See also: Report of Population Health Survey 2020-22 (Part II) (2023), Non-Communicable Diseases Watch, , Centre for Health Protection, Department of Health, HKSAR — https://www.chp.gov.hk/en/resources/29/283.html
- See also: Consequences of obesity, CDC (Centers for Disease Control and Prevention). — https://www.cdc.gov/obesity/basics/consequences.html